CLINICAL TRIAL: NCT04584489
Title: Prevalence and Incidence of Iron Deficiency in Cystic Fibrosis
Brief Title: Iron Metabolism in Cystic Fibrosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_0793
Record Dates: First submitted 2020-10-02; First posted 2020-10-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-08

CONDITIONS: Iron Metabolism, Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: iron stores assessment. — assessment of iron stores by measuring serum ferritin level (mandatory), serum iron and transferrin saturation.

SUMMARY:
Iron is a biologically essential micronutrient. Iron deficiency alters erythropoiesis and is considered as a major cause of disability worldwide. Interestingly, iron overload is never observed in cystic fibrosis contrarily to others chronic respiratory diseases. Moreover, iron deficiency reported prevalence in CF is very high (up to 60% in retrospective series) and is correlated to an alteration of respiratory function.

Cystic fibrosis patients should be tested annually for iron deficiency. Serum ferritin is the best diagnosis tool for iron deficiency (specificity 87% for a threshold < 30 µg/L). Previously published studies used less performant markers such as serum iron (< 12 µmol/L) or transferrin saturation (< 12%), which are markedly influenced by the systemic inflammation. CF patients experiences frequent pulmonary exacerbations leading to systemic inflammation: iron stores should therefore be assessed at optimal time with no inflammation.

The I-MUCO study aims to determine the exact prevalence of iron deficiency in CF patients. We aimed to identify risk factors for iron deficiency onset.

ELIGIBILITY:
Inclusion Criteria:

* Cystic fibrosis genetically proven.
* Age ≥ 18 years
* Systematic annual follow-up.

Exclusion Criteria:

* Dietary or drugs iron supplements
* Systemic inflammation or pulmonary exacerbation
* Lung transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: consecutive patients followed at the referral center for cystic fibrosis of Lyon (France).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-02-01 (Estimated); Study Completion 2021-02-01 (Estimated)

PRIMARY OUTCOMES:
prevalence of iron deficiency defined by serum ferritin ≤ 30 µg/L without inflammatory syndrome (C-reactive protein < 5 mg/L). | 1 year
  from inclusion to first documented up to 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de Ressources et de Compétences de la Mucoviscidose adulte de Lyon - Centre Hospitalier Lyon Sud, Pierre-Bénite, France